CLINICAL TRIAL: NCT03012646
Title: A Prospective, Multicenter, Single-arm Study to Evaluate the Safety and Tolerability of Inhaled Treprostinil in Subjects With Pulmonary Hypertension Due to Chronic Obstructive Pulmonary Disease
Brief Title: Safety and Tolerability of Inhaled Treprostinil in Adult PH Due to COPD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIN-PH-203
Record Dates: First submitted 2016-12-22; First posted 2017-01-06 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease
Keywords: Treprostinil; PH; COPD; 6 Minute Walk Test
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Inhaled Treprostinil (Experimental): Active Treprostinil for inhalation solution (0.6 mg/mL) delivered via an ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath.
  Interventions: Drug: Inhaled Treprostinil

INTERVENTIONS:
Drug: Inhaled Treprostinil — Inhaled treprostinil (6 mcg/breath) administered four times daily
  Other Names: Tyvaso

SUMMARY:
This is a multicenter, single-arm trial to evaluate the safety and efficacy of inhaled treprostinil in subjects with pre-capillary pulmonary hypertension (PH) associated with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of WHO Group 3 PH associated with COPD
2. Subjects are required to have a right heart catheterization (RHC) within one year prior to the first dose of study drug with the following parameters:

   1. Pulmonary vascular resistance (PVR) ≥ 4 Wood Units (WU) and
   2. A left ventricular end diastolic pressure (LVEDP) or pulmonary capillary wedge pressure (PCWP) of ≤ 12 mmHg if PVR ≥ 4 WU to < 6.25 WU or ≤ 15 mmHg if PVR ≥ 6.25 WU and
   3. A mean pulmonary arterial pressure (mPAP) of ≥ 30 mmHg
3. Clinical Diagnosis of COPD will be made using accepted Global Initiative for Chronic Obstructive Lung Disease (GOLD) diagnostic criteria, including Baseline spirometry with the following documented parameters:

   1. FEV1 < 65% predicted, and
   2. FEV1/ FVC < 70
4. Baseline 6MWD ≥ 100 meters

Exclusion criteria:

1. The subject has a diagnosis of pulmonary arterial hypertension (PAH) or PH for reasons other than COPD as outlined in inclusion criterion 3. This would include, but is not limited to, the concomitant presence of thromboembolic disease (acute or chronic), untreated or inadequately treated obstructive sleep apnea, connective tissue disease (including but not limited to systemic sclerosis/scleroderma, or systemic lupus erythematosus), sarcoidosis, interstitial lung disease,human immunodeficiency virus-1 infection, and other conditions under WHO Group 1, 2, 4, and 5 classifications.
2. The subject has received any Food and Drug Administration (FDA)-approved medication for the treatment of PAH (ie, prostacyclin, prostacyclin receptor agonist, endothelin receptor antagonist [ERA], phosphodiesterase type 5 inhibitor [PDE5-I],or soluble guanylate cyclase [sGC] stimulator) within 60 days of the first dose of study drug, except for acute vasoreactivity testing.
3. The subject has evidence of clinically significant left-sided heart disease as defined by the following criteria per the most recent assessment:

   1. Left ventricular end diastolic pressure (LVEDP) or pulmonary capillary wedge pressure (PCWP) >15 mmHg (or >12 mmHg if pulmonary vascular resistance [PVR] ≥4 to <6.25 WU)
   2. Left ventricular ejection fraction <40% as assessed by either angiography or echocardiography.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Among Participants through 48 Weeks | 48 weeks
  The incidence of adverse events among participants throughout the 48-week study will be measured by the number of participants analyzed and the percentage of those participants who experienced an adverse event.

SECONDARY OUTCOMES:
Change in 6-minute Walk Distance (6MWD) from Baseline to Week 48 | Baseline and Week 48
Change in plasma concentration of N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) from Baseline to Week 48 | Baseline and Week 48
Change in Forced Expiratory Volume (FEV1) in One Second from Baseline to Week 48 | Baseline and Week 48
Change in Forced Vital Capacity (FVC) from Baseline to Week 48 | Baseline and Week 48
Change in Lung Diffusion Capacity (DLCO) from Baseline to Week 48 | Baseline and Week 48
Change in right ventricular ejection fraction (RVEF) as assessed via cMRI from Baseline to Week 48 | Baseline and Week 48